CLINICAL TRIAL: NCT02208258
Title: Efficacy, Safety, and Performance Study of a Novel Device Designed to Manage Fecal Incontinence in Hospitalized Bedridden Patients With Liquid to Semi-formed Stool.
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Hospital had initiated a conflicting study, hence the study was terminated.
Sponsor: Consure Medical Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CON/2013/FI003
Record Dates: First submitted 2014-08-01; First posted 2014-08-05 (Estimated); Last update posted 2016-01-29 (Estimated); Status verified 2016-01

CONDITIONS: Fecal Incontinence
Keywords: fecal incontinence, consure medical, semi formed stool, stool management system
MeSH Terms: conditions — Fecal Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Consure 120 Stool Management System — Novel device designed to manage fecal incontinence in hospitalized bedridden patients with liquid to semi-formed stool.
  Other Names: Consure 120 SMS

SUMMARY:
The purpose of this study is to evaluate the safety, efficacy, and functionality of the Consure 120 Stool Management System in hospitalized bedridden patients suffering from fecal incontinence.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients, more than 18 years of age incontinent with liquid to semi-formed stool.
* Non-ambulatory, hospitalized patients.
* History of passage of at least 1 stool in 24 hours.

Exclusion Criteria:

* Patients with suspected or confirmed rectal mucosal impairment or pathology.
* Patients with have undergone descending colon or rectal surgery within the preceding six months.
* Patients with significant hemorrhoids, growth, fissure, stricture, stenosis or local pathology (either benign and malignant) as observed during rectal examination.
* Patients suspected to have impacted stool or is suffering from constipation.
* Patients with confirmed pregnancy or suspected to be pregnant.
* Patients that have planned MRI examination over the duration of the study.
* Patients who have suffered recent cardiac arrest within the preceding 3 months.
* Patients enrolled in another clinical study or clinical trial.
* Patients on oral or IV anti-coagulation (e.g., IV heparin drip, acetylsalicylic acid , Plavix). Subcutaneous heparin or low molecular weight heparin are acceptable).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-09; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Visual confirmation that fecal material is diverted into the external collection bag through the device. | 120 +/- 8 hours
  Yes or No response to visual observation of stool being collected through the transit sheath and collection bag.
Visual confirmation of no soiling, leaking or seepage of fecal secretions from the periphery of the device. | 120 +/- 8 hours
  Yes or No response to visual observation of soiling, leaking or seepage around periphery of device.
Number of hours for which the device stays on without change or removal. | 120 +/- 8 hours
  Quantitative measure of duration of device use. The cause of the change or removal will be documented.

SECONDARY OUTCOMES:
Visual confirmation of no active bleeding on the external periphery of the device (transit sheath or collection bag) over the usage of the device. | 120 +/- 8 hours
  Yes or No response from visual observation of any bleeding on the external periphery of the device.

CONTACTS AND LOCATIONS:
Locations (1):
- Sharp HealthCare, San Diego, California, United States